CLINICAL TRIAL: NCT06876233
Title: Mobile Cued Adherence Therapy (mCAT): A Scalable Habit Formation Intervention to Improve Blood Pressure Medication Adherence Based on a Widely Used Smartphone App
Brief Title: Mobile Cued Adherence Therapy (mCAT) for Blood Pressure Medication
Acronym: mCAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chad Stecher@asu.edu (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Wellth Inc. (Industry); Arizona State University (Other)
Responsible Party: Sponsor-Investigator, Chad Stecher@asu.edu, Assistant Professor, Arizona State University
Organization: Arizona State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00020282; R01HL171706 (NIH)
Record Dates: First submitted 2025-03-13; First posted 2025-03-14 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Medication Adherence; Hypertension; Habits
Keywords: habits; medication adherence; hypertension; blood pressure; mobile app
MeSH Terms: conditions — Medication Adherence; Hypertension; Habits

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Control participants will receive SMS reminders of each assessment point and monthly two-way SMS messages to provide AH pill-taking tips and to ask if participants are feeling dizziness or other symptoms of low blood pressure. Participants in the control group will not receive additional adherence reminders, financial incentives, or the Wellth app during the 24-month study.
- Wellth only (Experimental): Participants in the Wellth only group will receive daily financial incentives during the 4-month intervention for providing photo evidence of their pill taking using the mobile app Wellth (i.e. taking a daily picture of their pills in their hand and submitting it through the Wellth app). The Wellth app will also provide reminders at the end of the day if participants have not yet completed their daily check-in. Participants will also receive SMS reminders of each assessment point and monthly two-way SMS messages to provide AH pill-taking tips and to ask if participants are feeling dizziness or other symptoms of low blood pressure.
  Interventions: Behavioral: Wellth App
- Wellth + Cue (Experimental): Participants in the Wellth+Cue group will receive daily financial incentives during the 4-month intervention for providing photo evidence of their pill taking using the mobile app Wellth (i.e. taking a daily picture of their pills in their hand and submitting it through the Wellth app), conditional on using their action plan. The Wellth app will also provide reminders at the end of the day if participants have not yet completed their daily check-in. Participants will also receive SMS reminders of each assessment point and monthly two-way SMS messages to provide AH pill-taking tips and to ask if participants are feeling dizziness or other symptoms of low blood pressure.
  Interventions: Behavioral: Action Planning; Behavioral: Wellth + Cue

INTERVENTIONS:
Behavioral: Wellth App — Participants will be eligible to receive $30 at the end of four consecutive 30-day periods ($120 in total) if they demonstrate complete medication adherence through the Wellth app (i.e. taking a daily picture of their pills in their hand and submitting it through the Wellth app). Photos must be submitted within a 2-hour window around a specific time of day chosen by the participant and set at the start of each 30-day period. They will lose $2 (from their $30 total) for every day they miss a medication check-in within their pre-set 2-hour window with the Wellth app. The Wellth app will also provide reminders at the end of the day if participants have not yet completed their daily check-in.
  Arms: Wellth only
Behavioral: Action Planning — Participants will learn about habits and the importance of contextual cues for triggering their AH pill taking, and be asked to complete an electronic worksheet with a detailed description of their personalized contextual cue in terms of its: 1) location (e.g., where in the participant's house or office does this cue occur); 2) time of day; 3) preceding action (e.g., "I usually go to the bathroom before making coffee"); and 4) a visual cue (e.g., "my coffee cup will trigger pill taking").
  Arms: Wellth + Cue
Behavioral: Wellth + Cue — Participants will be eligible to receive $30 at the end of four consecutive 30-day periods ($120 in total) if they submit daily evidence of their medication adherence habit using the Wellth app (i.e. one photo that provides evidence of pill-taking and one photo that provides evidence of their contextual cue, which participants will select and specify on their comprehension survey at the start of the study). Photos must be submitted within a 2-hour window around a specific time of day chosen by the participant and set at the start of each 30-day period. They will lose $2 (from their $30 total) for every day they miss a medication check-in (plus evidence of their contextual cue) within their pre-set 2-hour window with the Wellth app. The Wellth app will also provide reminders at the end of the day if participants have not yet completed their daily check-in.
  Arms: Wellth + Cue

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of a novel mobile health-based habit formation intervention for increasing and maintaining adherence to anti-hypertensive (AH) medication among people living with hypertension and indicate medication nonadherence. The main questions it aims to answer are:

* Can daily incentives for AH pill taking increase and maintain AH medication adherence, control blood pressure, and reduce healthcare utilization and costs?
* Can daily incentives for AH pill taking, combined with action planning (e.g., "After I drink my morning coffee, I will take my medication.") increase and maintain medication adherence, control blood pressure, and reduce healthcare utilization and costs?
* What aspects of daily incentives and/or action planning do participants find most helpful or effective for AH medication adherence?
* What barriers exist for participants who receive daily incentives and/or action planning?

Researchers will compare three study groups: those who only receive daily incentives for the AH pill taking, those who receive daily incentives for AH pill taking combined with action planning, and a control group (who do not receive daily incentives for AH pill taking or action planning). By comparing these three groups, the researchers will be able to determine the effectiveness of the daily incentives with or without action planning for promoting long-term AH medication adherence, reduce healthcare costs, and improve blood pressure.

Participants will:

* Complete 5 online surveys over the course of 2 years (baseline, month 4, month 8, month 12, month 24).
* Submit blood pressure reading for 7 consecutive days after each survey timepoint.
* Submit photo evidence of their AH pill taking for 4 months (intervention groups only).

The highest- and lowest-performing participants in each intervention group will also be invited to complete a 30-minute interview to identify additional factors that contributed to either successful or unsuccessful completion of the intervention.

ELIGIBILITY:
Eligibility Criteria:

* Aged 18 years or older
* Currently diagnosed with hypertension (either stage I or stage II hypertension)
* Able to read/write/understand English
* Have daily access to a smartphone
* Engaged in hypertension care: Already been prescribed hypertension medication for a minimum of 12 months at the time of study enrollment
* Demonstrated AH medication nonadherence by having over 73 days without documented AH medication prescription coverage (observable in Arizona Health Care Cost Containment System (AHCCCS) prescription drugs claims) in the past 12 months (i.e. <80% mean adherence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | 24 months prior to the study through the 24-month study period
  The investigators will use Medicaid's prescription data to construct the Primary Outcome of AH medication adherence using the date and supply of pills for each new prescription or refill to determine the number of days in a month a client had pills available. Since refills are often made before an existing prescription ends, the supply of new medications will be counted on days following the last available dose of the prior prescription. The number of days with available AH medication(s) will be divided by the total number of days in the same month to calculate the proportion of days covered (PDC), which will range from 0 and 1.
Cardiovascular Health | Baseline, after the 4-month intervention, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  All participants will be asked to submit blood pressure readings for seven consecutive days after baseline activities, and be reminded via SMS and email to submit readings after the 4-month intervention and again after the month 8, 12, and 24 assessments. The investigators will calculate the Primary Outcome measure of blood pressure as participants' mean and coefficient of variation in systolic and diastolic blood pressure over the seven-day interval.

SECONDARY OUTCOMES:
Healthcare Utilization and Costs | 24 months prior to the study through the 24-month study period
  The investigators will use Medicaid's encounters and reimbursement costs data to construct our Secondary Outcomes of healthcare utilization and costs. The investigators will generate separate monthly measures of the number of unique encounters, as well as the number of days in an emergency department, and inpatient and outpatient healthcare settings. Since a single encounter can be billed multiple times (thus appearing multiple times in the data) or last multiple days, the investigators will remove duplicate encounter claims based on the date of service, diagnostic codes, and procedure costs associated with each encounter. The investigators will separately measure the monthly AHCCCS reimbursement costs for all unique encounters in each healthcare setting.

OTHER OUTCOMES:
Self-Reported Habit Strength | Baseline, after the 4-month intervention, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Habit strength (i.e., behavioral automaticity) will be measured using the Self-Reported Behavioral Automaticity Index (SRBAI), a frequently used 4-item subscale of the Self-Reported Habit Index (SRHI). The SRBAI assesses the degree to which a given behavior (e.g., pill taking) is an automatic or unconscious process. Scores range from 5-20, with higher scores indicating greater self-reported habit strength
Wellth-measured Habit Strength | Continuously during 24-month study period
  This is an objective measure of habit strength that will provide an estimate of the monthly proportion of days with cued pill-taking. Specifically, the investigators will estimate the monthly proportion of days with a valid cue check-in (i.e., containing photographic evidence of a participant's contextual cue) that is successfully submitted within +/- 1 hour of the stated time when the participant's cue occurs during the day. This proportion will range from 0 to 1, where a higher proportion indicates greater habit strength.
Present Bias | Baseline, after the 4-month intervention, 8-month follow-up, 12-month follow-up, and 24-month follow-up
  Present bias (i.e., the tendency for monetary rewards now to be valued higher relative to those at any future point) will be measured using the Multiple Price List Task, which asks participants to choose between smaller rewards received sooner and larger rewards received later. This is estimated by comparing participants' willingness to forego rewards received today versus future periods, relative to their willingness to forego rewards received in two weeks versus points after two weeks. A person's willingness to forego rewards today relative to forgoing rewards in two weeks for future rewards indicates their degree of present bias.

CONTACTS AND LOCATIONS:
Locations (1):
- Wellth Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers. Aggregated data will be available upon request.